CLINICAL TRIAL: NCT03155087
Title: The Influence of AMPK Subunit Alpha (PRKAA2) Genetic Polymorphisms With Susceptibility to Chinese Type 2 Diabetes Mellitus and Diabetic Nephropathy
Brief Title: PRKAA2 Genetic Polymorphisms and Its Susceptibility to Chinese Type 2 Diabetes Mellitus and Diabetic Nephropathy
Status: Completed | Type: Observational
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zhi Li, Principal Investigator, People's Hospital of Zhengzhou University
Other Study IDs: 2016ys5
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
Keywords: T2DM; genetic polymorphism; diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T2DM patients: Metformin dosages ranged from 500 to 2000 mg per day
  Interventions: Drug: Metformin
- healthy subjects: the healthy subjects was not intervened

INTERVENTIONS:
Drug: Metformin
  Groups: T2DM patients

SUMMARY:
Metformin is a classical oral antidiabetic drug, often recommended to be the first-choice treatment of type 2 diabetes mellitus (T2DM). Based on the previous research on PRKAA2, STK11 and diabetes, this study aimed to investigate the distributive characteristic of PRKAA2 and STK11 polymorphisms and the potential influence of STK11polymorphisms on metformin efficacy among Chinese T2DM patients, discuss the association of PRKAA2 polymorphisms between T2DM patients and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T2DM in keeping with the WHO criteria in 1999 [14], with fasting blood glucose (FBG) ≥ 7.0mmol ⁄ L and ⁄ or postprandial blood glucose (PBG) ≥ 11.1mmol ⁄ L; not using other antidiabetic drugs within the experimental period.

Exclusion Criteria:

* other significant illness such as cancer, myocardial infarction, stroke, severe liver, and kidney disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study recruited 500 T2DM patients and 250 healthy subjects who meet the enrollment cirterion from Zhengzhou Central Hospital during the period of July 2013 to December 2015 randomly.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the incidence of T2DM | Jan 2014-Dec 2015
  people whose fasting plasma glucose ≥7.0 mmol/L and/or postprandial plasma glucose ≥11.1 mmol/L is diagnosed with T2DM.

SECONDARY OUTCOMES:
metformin efficacy----the decrease level of HbA1c | Jan 2014-Dec 2015
  patients whose HbA1c levels is decreased by more than 0.5 % from the baseline is deemed as the response group, while the decrease in HbA1c levels less than 0.5 % from the baseline is deemed as the non-response group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Q, Li C, Li H, Zeng L, Kang Z, Mao Y, Tang X, Zheng P, He L, Luo F, Li Z. STK11 rs2075604 Polymorphism Is Associated with Metformin Efficacy in Chinese Type 2 Diabetes Mellitus. Int J Endocrinol. 2017;2017:3402808. doi: 10.1155/2017/3402808. Epub 2017 Jul 9. PMID 28775741